CLINICAL TRIAL: NCT03021486
Title: Haloperidol and/or Chlorpromazine for Refractory Agitated Delirium in the Palliative Care Unit
Brief Title: Haloperidol With or Without Chlorpromazine in Treating Delirium in Patients With Advanced, Metastatic, or Recurrent Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2016-0687; NCI-2017-01065 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0687 (Other: M D Anderson Cancer Center); R21NR016736 (NIH)
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2022-09-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Neoplasm; Delirium; Locally Advanced Malignant Neoplasm; Metastatic Malignant Neoplasm; Recurrent Malignant Neoplasm
MeSH Terms: conditions — Delirium; Neoplasm Metastasis; Recurrence | interventions — Chlorpromazine; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I (haloperidol) (Experimental): Patients receive haloperidol IV over 3-15 minutes every 4 hours in the absence of unacceptable toxicity.
  Interventions: Drug: Haloperidol; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (chlorpromazine) (Experimental): Patients receive chlorpromazine IV over 3-15 minutes every 4 hours in the absence of unacceptable toxicity.
  Interventions: Drug: Chlorpromazine; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (haloperidol, chlorpromazine) (Experimental): Patients receive haloperidol and chlorpromazine IV over 3-15 minutes every 4 hours in the absence of unacceptable toxicity.
  Interventions: Drug: Chlorpromazine; Drug: Haloperidol; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Chlorpromazine — Given IV
  Other Names: Chlor-PZ; Thorazine
  Arms: Group II (chlorpromazine); Group III (haloperidol, chlorpromazine)
Drug: Haloperidol — Given IV
  Other Names: Haldol; McN-JR-1625; R 1625; R-1625
  Arms: Group I (haloperidol); Group III (haloperidol, chlorpromazine)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II/III trial studies how well haloperidol with or without chlorpromazine works in treating delirium in patients with cancer that has spread to other parts of the body or has come back. Haloperidol and chlorpromazine may control the symptoms of delirium (loss of contact with reality) in patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the within-arm effect of haloperidol dose escalation, rotation to chlorpromazine, and combination therapy on agitation intensity (Richmond Agitation Sedation Scale [RASS]) over 24 hours in patients admitted to an acute palliative care unit (APCU) who did not experience a response to low-dose haloperidol.

SECONDARY OBJECTIVES:

I. Obtain preliminary estimates of the effects of haloperidol dose escalation, rotation to chlorpromazine, and combination therapy on (1) the proportion of patients with target RASS -2 to 0, (2) delirium-related distress in nurses and caregivers (delirium experience questionnaire), (3) symptom expression (Edmonton Symptom Assessment Scale), (4) delirium severity (Memorial Delirium Assessment Scale), (5) the need for neuroleptics, (6) delirium recall (Delirium Recall Questionnaire), (7) adverse effects and (8) quality of end-of-life (Quality of Death and Dying questionnaire) over time.

II. Obtain preliminary estimates of the between-arm effect size among haloperidol dose escalation, rotation to chlorpromazine, and combination therapy in the first 24 hours.

III. To assess caregiver and nurse preferences regarding proxy sedation goals. IV. To examine the feasibility of novel measures for the assessment of agitation with continuous video monitoring.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I: Patients receive haloperidol intravenously (IV) over 3-15 minutes every 4 hours in the absence of unacceptable toxicity.

GROUP II: Patients receive chlorpromazine IV over 3-15 minutes every 4 hours in the absence of unacceptable toxicity.

GROUP III: Patients receive haloperidol and chlorpromazine IV over 3-15 minutes every 4 hours in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion:

1. [Patients] Diagnosis of advanced cancer (defined as locally advanced, metastatic recurrent, or incurable disease)
2. [Patients] Admitted to the acute palliative care unit
3. [Patients] Delirium as per DSM-V criteria (The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5))
4. [Patients] Hyperactive or mixed delirium with RASS >/=1 in the past 24 h (RASS>/=+1 indicates any degree of restlessness. In the electronic medical record nursing note, this behavior would be indicated by any documentation of "restless", "agitated", "hyperactive", "pulling on devices/IV" or similar wording).
5. [Patients] On scheduled haloperidol for delirium (</=8 mg in the past 24 h) or rescue haloperidol of >/=4 mg for restlessness/agitation in the past 24 h
6. [Patients] Age 18 years or older
7. [Family Caregivers] Patient's spouse, adult child, sibling, parent, other relative, or significant other (defined by the patient as a partner)
8. [Family Caregivers] Age 18 years or older

Exclusion:

1. [Patients] History of myasthenia gravis or acute narrow angle glaucoma
2. [Patients] History of neuroleptic malignant syndrome or active seizure disorder (with seizure episode within the past week)
3. [Patients] History of Parkinson's disease or Alzheimer's dementia
4. [Patients] History of prolonged QTc interval (>500 ms) if documented by ECG within the past month
5. [Patients] History of hypersensitivity to haloperidol or chlorpromazine
6. [Patients] On scheduled chlorpromazine within the past 48 h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2027-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hui D, De La Rosa A, Wilson A, Nguyen T, Wu J, Delgado-Guay M, Azhar A, Arthur J, Epner D, Haider A, De La Cruz M, Heung Y, Tanco K, Dalal S, Reddy A, Williams J, Amin S, Armstrong TS, Breitbart W, Bruera E. Neuroleptic strategies for terminal agitation in patients with cancer and delirium at an acute palliative care unit: a single-centre, double-blind, parallel-group, randomised trial. Lancet Oncol. 2020 Jul;21(7):989-998. doi: 10.1016/S1470-2045(20)30307-7. Epub 2020 May 29. PMID 32479786
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants (age>18) with an active diagnosis of cancer were recruited between palliative and supportive Care unit at MD Anderson Cancer Center who met the inclusion and exclusion criteria.
Pre-assignment Details: A total of 70 participants were consented, 2 were inevaluable and 68 were randomly assigned for interventions.
Groups:
- Escalation Group: Participants receive 2 mg of haloperidol IV over 3-15 minutes every 4 hours in absence of unacceptable toxicity.
- Rotation Group: Participants receive 25 mg of chlorpromazine IV over 3-15 minutes every 4 hours in the absence of unacceptable toxicity.
- Combination Group: Participants receive 1 mg of haloperidol and 12.5 mg of chlorpromazine IV over 3-15 minutes every 4 hours in the absence of unacceptable toxicity.
Period: Overall Study
Arm/Group | Escalation Group | Rotation Group | Combination Group
Started | 23 | 22 | 23
Completed | 15 | 16 | 14
Not Completed | 8 | 6 | 9
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Did not develop an RASS score of at least >= 1 | 7 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escalation Group | Rotation Group | Combination Group | Total
Number analyzed (Participants) | 15 | 16 | 14 | 45
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [61 to 75] | 63 [59 to 70] | 60 [57 to 74] | 64 [58 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 8 | 19
  Male | 10 | 10 | 6 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 14 | 15 | 12 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 11 | 14 | 12 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 14 | 45
Education [Count of Participants; unit: Participants]
  Some High school or less | 1 | 0 | 3 | 4
  Completed High School | 5 | 7 | 4 | 16
  Some College | 4 | 3 | 3 | 10
  College | 4 | 5 | 2 | 11
  Advanced degree | 1 | 1 | 2 | 4
Cancer Type [Count of Participants; unit: Participants]
  Breast | 3 | 1 | 1 | 5
  Genitourinary | 1 | 1 | 2 | 4
  Gastrointestinal | 5 | 7 | 2 | 14
  Gynecological | 0 | 0 | 1 | 1
  Hematological | 0 | 3 | 2 | 5
  Respiratory | 4 | 3 | 3 | 10
  Others | 2 | 1 | 3 | 6
Metastatic cancer or advanced stage disease [Count of Participants; unit: Participants] | 15 | 16 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Richmond Agitation Sedation Score (RASS) (0-24h)
Description: RASS score is a 10-point scale with scores ranging from +4 (very combative, violent) to -5 (unarousable). The primary outcome was mean change in RASS score between time 0 (immediately before initiation of masked treatment) and 24 h later. The Richmond Agitation-Sedation Scale (RASS) was developed by a multidisciplinary team at Virginia Commonwealth University in Richmond; it is a validated method used to avoid oversedation in the Intensive Care Unit.
Time Frame: Time 0 or Baseline and 24 hours after study medication administration
Population: Analysis included 31 participants who completed 24 hours of the study.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 10 | 11 | 10
score on a scale | -3.6 [-5.0 to -2.2] | -3.3 [-4.4 to -2.2] | -3.0 [-4.6 to -1.4]
Statistical Analysis 1: Comparison: Escalation Group vs Rotation Group vs Combination Group; Test type: Other; p = 0.71, Wilcoxon Rank Sum Test

2. Secondary Outcome: Percentage of Participants With RASS Score -2 to 0
Description: RASS score is a 10-point scale with scores ranging from +4 (very combative, violent) to -5 (unarousable). The Secondary outcome was the percentage of participants with target RASS score of -2 to 0 within the first 24 hours. The Richmond Agitation-Sedation Scale (RASS) was developed by a multidisciplinary team at Virginia Commonwealth University in Richmond; it is a validated method used to avoid over sedation in the Intensive Care Unit.
Time Frame: Time 0 or Baseline and 24 hours later.
Population: Analysis included 31 participants who completed 24 hours of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Combination Group: Participants receive 1 mg of haloperidol and 12·5 mg of chlorpromazine IV over 3-15 minutes every 4 hours in the absence of unacceptable toxicity.
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 10 | 11 | 10
Participants | 2 | 3 | 5

3. Secondary Outcome: Change in RASS Score (0-30 Minutes)
Description: RASS score is a 10-point scale with scores ranging from +4 (very combative, violent) to -5 (unarousable). The secondary outcome was mean change in RASS score between time 0 (immediately before initiation of masked treatment) and 30 minutes later. The Richmond Agitation-Sedation Scale (RASS) was developed by a multidisciplinary team at Virginia Commonwealth University in Richmond; it is a validated method used to avoid over sedation in the Intensive Care Unit.
Time Frame: Time 0 or Baseline and 30 minutes later.
Population: Analysis included 45 participants who completed first 30 minutes of study
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 15 | 16 | 14
score on a scale | -2.6 [-3.6 to -1.6] | -2.4 [-3.0 to -1.8] | -2.1 [-3.0 to -1.3]
Statistical Analysis 1: Comparison: Escalation Group vs Rotation Group vs Combination Group; Test type: Other; p = 0.86, Wilcoxon Rank Sum Test

4. Secondary Outcome: Number of Participants With RASS Score of >=1
Description: RASS score is a 10-point scale with scores ranging from +4 (very combative, violent) to -5 (unarousable). The secondary outcome was the proportion of breakthrough restlessness participants with a RASS score of >=1 during the first 24 hours. The Richmond Agitation-Sedation Scale (RASS) was developed by a multidisciplinary team at Virginia Commonwealth University in Richmond; it is a validated method used to avoid oversedation in the Intensive Care Unit.
Time Frame: 0 or Baseline and 24 hours later
Population: Analysis included 45 participants who completed first 24 hours of study
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 15 | 16 | 14
Participants | 12 | 7 | 9
Statistical Analysis 1: Comparison: Escalation Group vs Rotation Group vs Combination Group; Test type: Other; p = 0.12, Two-tailed Fisher's exact test

5. Secondary Outcome: Pattern of Medication Use
Description: Use of neuroleptics and benzodiazepines during the first 24 hours was retrieved from the Medication Administration Record.
Time Frame: Baseline and 24 hours
Population: Analysis included 45 participants who were still on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 15 | 16 | 14
Participants
  Need for study med dose escalation in first 24 hrs | 4 | 1 | 7
  Benzodiazepine use in first 24 hrs (scheduled) | 1 | 0 | 0
  Benzodiazepine use in first 24 hrs (as needed) | 0 | 0 | 4
Statistical Analysis 1: Comparison: Escalation Group vs Rotation Group vs Combination Group; Test type: Other; p = 0.007, Two-tailed Fisher's exact test

6. Secondary Outcome: Perceived Comfort Level as Assessed by Caregiver
Description: On day 1 (after initiation of blinded treatment), we asked the blinded caregivers to provide their overall impression of change in patient comfort level and the agitation level. The response ranged from "strongly agree", "agree", "neutral", "disagree", and "strongly disagree". In this study, "strongly agree" and "agree" were combined for analysis. The participants who reported 'Agree' and 'Strongly Agree' responses to perceived comfort level have a high level of comfort (more comfortable). And similarly, the participants who reported 'Agree' and 'Strongly Agree' responses to perceived agitation level have a low level of agitation (less agitated).
Time Frame: Baseline and 24 hour
Population: Analysis included 37 participants who completed this questionnaire at that time point
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 13 | 14 | 10
Participants
  Perceived To Have A High Level of Comfort (More Comfortable) | 8 | 10 | 6
  Perceived To Have A Low Level of Agitation (Less Agitated) | 9 | 10 | 6
Statistical Analysis 1: Comparison: Escalation Group vs Rotation Group vs Combination Group; Perceived Comfort level as assessed by caregiver; Test type: Other; p = 0.83, Two-tailed Fisher's exact test
Statistical Analysis 2: Comparison: Escalation Group vs Rotation Group vs Combination Group; Perceived agitation level as assessed by caregiver; Test type: Other; p = 0.82, Two-tailed Fisher's exact test

7. Secondary Outcome: Perceived Comfort Level as Assessed by Nurse
Description: as for outcome 6
Time Frame: Baseline and 24 hour
Population: Analysis included 37 participants who completed this questionnaire at that time point
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 14 | 12 | 11
Participants
  Perceived To Have A High Level of Comfort (More Comfortable) | 9 | 9 | 7
  Perceived To Have A Low Level of Agitation (Less Agitated) | 8 | 8 | 7
Statistical Analysis 1: Comparison: Escalation Group vs Rotation Group vs Combination Group; Perceived Comfort level as assessed by nurse; Test type: Other; p = 0.82, Two-tailed Fisher's exact test
Statistical Analysis 2: Comparison: Escalation Group vs Rotation Group vs Combination Group; Perceived agitation level as assessed by nurse; Test type: Other; p = 0.91, Two-tailed Fisher's exact test

8. Secondary Outcome: Change in Delirium Experience Questionnaire
Description: This 14-item questionnaire examines both the recalled frequency of 7 delirium symptoms and associated distress in the rater: disorientation to time, disorientation to place, visual hallucinations, tactile hallucinations, auditory hallucinations, delusional thoughts and psychomotor agitation. The score for recalled frequency ranges between 0 and 4, where 0=not present, 1=a little of the time, 2=some of the time, 3=good part of the time, and 4=most or all of the time. The score for distress in the rater related to each delirium symptom also ranges from 0 to 4, where 0=no distress, 1=a little, 2=a fair amount, 3=very much and 4=extremely distressed. Due to an error in the data collection form, the last category was omitted as a choice and thus the score only ranged from 0 to 3.
Time Frame: Baseline and Day 3
Population: Analysis included 37 participants who completed this questionnaire at that time point.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 14 | 12 | 11
score on a scale
  Nursing assessment, disorientation to time - frequency | -0.8 [-1.7 to 0.1] | -0.8 [-1.6 to 0.1] | 0.2 [-0.8 to 1.1]
  Nursing assessment, disorientation to place - frequency | -0.9 [-1.7 to -0.1] | -0.8 [-1.7 to 0.2] | 0.3 [-0.7 to 1.3]
  Nursing assessment, visual hallucination - frequency | -1 [-1.6 to -0.5] | 0 [-0.6 to 0.6] | -0.7 [-1.5 to 0]
  Nursing assessment, tactile hallucination - frequency | -0.4 [-1.1 to 0.3] | 0.1 [-0.1 to 0.3] | -0.9 [-1.7 to -0.2]
  Nursing assessment, auditory hallucination - frequency | -0.1 [-0.5 to 0.2] | 0.1 [-0.1 to 0.3] | -0.4 [-0.8 to 0.1]
  Nursing assessment, delusional thoughts - frequency | -0.8 [-1.5 to 0] | 0 [-0.3 to 0.3] | 0.2 [-0.5 to 0.9]
  Nursing assessment, psychomotor agitation- frequency | -1.2 [-1.9 to -0.5] | -0.8 [-1.7 to 0] | -0.4 [-1 to 0.3]
  Nursing assessment, disorientation to time - distress | -0.3 [-0.6 to 0.1] | -0.3 [-0.7 to 0.2] | -0.5 [-1.2 to 0.2]
  Nursing assessment, disorientation to place - distress | -0.3 [-0.6 to 0.1] | -0.3 [-0.7 to 0.2] | -0.4 [-1.1 to 0.4]
  Nursing assessment, visual hallucination - distress | -0.6 [-1.3 to 0] | 0.1 [-0.1 to 0.3] | -0.4 [-0.9 to 0.2]
  Nursing assessment, tactile hallucination - distress | -0.5 [-1.1 to 0.1] | 0 [0 to 0] | -0.5 [-1.1 to 0.2]
  Nursing assessment, auditory hallucination - distress | -0.3 [-0.9 to 0.3] | 0 [0 to 0] | -0.2 [-0.6 to 0.2]
  Nursing assessment, delusional thoughts - distress | -0.6 [-1.4 to 0.1] | 0 [0 to 0] | -0.1 [-0.6 to 0.4]
  Nursing assessment, psychomotor agitation - distress | -0.8 [-1.4 to -0.2] | -0.5 [-0.9 to -0.1] | -0.8 [-1.5 to -0.1]
Statistical Analysis 1: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, disorientation to time - frequency; Test type: Other; p = 0.12, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, disorientation to place - frequency; Test type: Other; p = 0.07, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, visual hallucination - frequency; Test type: Other; p = 0.051, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, tactile hallucination - frequency; Test type: Other; p = 0.048, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, auditory hallucination - frequency; Test type: Other; p = 0.15, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, delusional thoughts - frequency; Test type: Other; p = 0.10, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, psychomotor agitation- frequency; Test type: Other; p = 0.15, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, disorientation to time - distress; Test type: Other; p = 0.98, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, disorientation to place - distress; Test type: Other; p = 0.93, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, visual hallucination - distress; Test type: Other; p = 0.08, Wilcoxon Rank Sum Test
Statistical Analysis 11: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, tactile hallucination - distress; Test type: Other; p = 0.28, Wilcoxon Rank Sum Test
Statistical Analysis 12: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, auditory hallucination - distress; Test type: Other; p = 0.83, Wilcoxon Rank Sum Test
Statistical Analysis 13: Comparison: Escalation Group vs Rotation Group; Nursing assessment, delusional thoughts - distress; Test type: Other; p = 0.22, Wilcoxon Rank Sum Test
Statistical Analysis 14: Comparison: Escalation Group vs Rotation Group vs Combination Group; Nursing assessment, psychomotor agitation - distress; Test type: Other; p = 0.75, Wilcoxon Rank Sum Test

9. Secondary Outcome: Memorial Delirium Assessment Scale (MDAS)
Description: The Memorial Delirium Assessment Scale (MDAS) is a 10-item clinician-rated assessment scale validated for assessment of delirium in cancer patients. It examines the level of consciousness, disorientation, memory, recall, attention, disorganized thinking, perceptual disturbance, delusions, psychomotor activity and sleep, assigning a score between 0 to 3, for a total score between 0-30. A total score of 13 or higher indicates delirium. We measured the change in Memorial Delirium Rating scale between baseline and 24 hours.
Time Frame: Baseline and 24 hours
Population: Analysis included 30 participants who completed this questionnaire at that time point
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 9 | 11 | 10
score on a scale | -2.7 [-6 to 0.7] | 1 [-0.3 to 2.3] | 0.3 [-2.9 to 3.5]
Statistical Analysis 1: Comparison: Escalation Group vs Rotation Group vs Combination Group; Test type: Other; p = 0.09, Wilcoxon Rank Sum Test

10. Secondary Outcome: Edmonton Expression Assessment System, ESAS
Description: Edmonton Symptom Assessment System (ESAS) has been validated and widely used in different clinical settings, including the acute palliative care unit. It assessed the average symptom intensity of 10 symptoms over the past 24 hours. Each symptom was assessed using an 11-point numeric rating scale, ranging from 0 (none) to 10 (worst). It was measured as change in ESAS as Perceived by Caregivers between baseline and day 1, mean.
Time Frame: Baseline and 24 hours
Population: Analysis included 33 participants who completed this questionnaire at that time point. Note that 9 participants completed 'feeling of well being' question for Combination group, and 13 participants completed 'pain' and 'sleep' questions for Escalation group
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 13 | 11 | 10
score on a scale
  Pain | -1.3 [-3.1 to 0.5] | -4.1 [-5.8 to -2.4] | -1.1 [-2.3 to 0.1]
  Fatigue: number analyzed (Participants) | 12 | 11 | 10
  Fatigue | -0.5 [-2.6 to 1.6] | -3 [-5.9 to -0.1] | 1 [-0.8 to 2.8]
  Nausea: number analyzed (Participants) | 12 | 11 | 10
  Nausea | 0.1 [-0.3 to 0.5] | -1.8 [-3.1 to -0.5] | -0.4 [-1.1 to 0.3]
  Depression: number analyzed (Participants) | 12 | 11 | 10
  Depression | -1.4 [-3.2 to 0.4] | -1.2 [-3.6 to 1.2] | -0.8 [-2.3 to 0.7]
  Anxiety: number analyzed (Participants) | 12 | 11 | 10
  Anxiety | -1.5 [-3.7 to 0.7] | -4.8 [-6.6 to -3.1] | -0.9 [-3.4 to 1.6]
  Drowsiness: number analyzed (Participants) | 12 | 11 | 10
  Drowsiness | -0.2 [-1.9 to 1.6] | -0.6 [-2.2 to 1.1] | 0.7 [-1.8 to 3.2]
  Appetite: number analyzed (Participants) | 12 | 11 | 10
  Appetite | -0.3 [-2 to 6.2] | -0.6 [-4 to 2.9] | 0.1 [-2.3 to 2.5]
  Feeling of well being*: number analyzed (Participants) | 12 | 11 | 9
  Feeling of well being* | 0.2 [-2 to 2.3] | -1.6 [-4.7 to 1.6] | 0 [-2.7 to 2.7]
  Shortness of breath: number analyzed (Participants) | 12 | 11 | 10
  Shortness of breath | 0.8 [0 to 1.6] | -2.2 [-5 to 0.6] | 0 [-1.7 to 1.7]
  Sleep | -2.7 [-4.7 to -0.7] | -5.1 [-7.3 to -2.9] | -2.7 [-4.5 to -0.9]
Statistical Analysis 1: Comparison: Escalation Group vs Rotation Group vs Combination Group; Mean change in pain; Test type: Other; p = 0.02, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Escalation Group vs Rotation Group vs Combination Group; Mean change in Fatigue; Test type: Other; p = 0.10, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Escalation Group vs Rotation Group vs Combination Group; Mean change in Nausea; Test type: Other; p = 0.02, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Escalation Group vs Rotation Group vs Combination Group; Mean change in Depression; Test type: Other; p = 0.97, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Escalation Group vs Rotation Group vs Combination Group; Mean change in Anxiety; Test type: Other; p = 0.03, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Escalation Group vs Rotation Group vs Combination Group; Mean change in Drowsiness; Test type: Other; p = 0.68, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Escalation Group vs Rotation Group vs Combination Group; Mean change in Appetite; Test type: Other; p = 0.80, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Escalation Group vs Rotation Group vs Combination Group; Mean change in Feeling of well being; Test type: Other; p = 0.45, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Escalation Group vs Rotation Group vs Combination Group; Mean change in Shortness of breath; Test type: Other; p = 0.16, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Escalation Group vs Rotation Group vs Combination Group; Mean change in Sleep; Test type: Other; p = 0.12, Wilcoxon Rank Sum Test

11. Secondary Outcome: Udvalg for Kliniske Undersogelser, UKU
Description: We also documented the selected adverse effects associated with neuroleptics using the Udvalg for Kliniske Undersogelser (UKU) side effects rating scale. Specifically, we assessed 8 neurologic symptoms (dystonia, rigidity, hypokinesia/akinesia, hyperkinesia, tremor, akathisia, epileptic seizures, paraesthesias). We are reporting only the neurologic symptoms (tremor and akathisia) that had changes during the study. Each item was assigned a score by the research coordinator 0 (absent) to 3 (most severe) based on symptom severity of the last 3 days.
Time Frame: Baseline and 3 days
Population: Analysis included 25 participants who were still on study
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Group | Rotation Group | Combination Group
Number analyzed (Participants) | 7 | 9 | 9
Participants
  Tremor (decreased) | 0 | 0 | 1
  Akathisia (decreased) | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline and 24 hr.
Groups:
- Escalation Group (Haloperidol Dose Escalation Group): Participants receive 2 mg of haloperidol IV over 3-15 minutes every 4 hours in absence of unacceptable toxicity.
Arm/Group | Escalation Group (Haloperidol Dose Escalation Group) | Rotation Group | Combination Group
All-Cause Mortality (participants affected / at risk) | 14/15 | 16/16 | 14/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 6/15 | 5/16 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation Group (Haloperidol Dose Escalation Group) (N=15) | Rotation Group (N=16) | Combination Group (N=14)
Akathisia (Nervous system disorders) | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Cardiac disorders) | 6 | 5 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT03021486/Prot_SAP_000.pdf